CLINICAL TRIAL: NCT04860531
Title: The Role of Intra-articular Injection of Autologous Platelet Rich Plasma Versus Corticosteriods in Treatment of Synovitis in Lumbar Facet Joint Disease
Brief Title: The Role of Intra-articular Injection of PRP Versus Corticosteriods in Treatment of Lumbar Facet Disease
Acronym: PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shahdan Yousry Abdelmonem Kotb, Assistant Lecturer of Physical medicine and Rehabilitation, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 222 / 2017
Record Dates: First submitted 2021-01-03; First posted 2021-04-27 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Lumbar Facet Joint Syndrome
Keywords: Platelet Rich Plasma
MeSH Terms: interventions — Lidocaine; Betamethasone

STUDY DESIGN:
Intervention Model Description: The participants are assigned for intra-articular injection of lumbar facet joint to either; Group (I) to be injected with autologous platelet rich plasma and Group (II) to be injected with corticosteroids(a mixture of 0.5% lidocaine and 5mg/ml of betamethasone) . The treated segments will be determined by clinical signs and MRI detected facet joint synovitis .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (I) Platelet Rich Plasma (Active Comparator): The participants are randomly assigned for intra-articular injection with autologous platelet rich plasma . The treated segments are determined by clinical signs and MRI detected facet joint synovitis .
  Interventions: Drug: Lumbar Facet Joints intra-articular injection with Platelet Rich Plasma
- Group (II) Corticosteroids (Active Comparator): The participants are randomly assigned for intra-articular injection with corticosteroids(a mixture of 0.5% lidocaine and 5mg/ml of betamethasone) . The treated segments will be determined by clinical signs and MRI detected facet joint synovitis .
  Interventions: Drug: Lumbar Facet Joints intra-articular injection with a mixture of 0.5% lidocaine and 5mg/ml of betamethasone

INTERVENTIONS:
Drug: Lumbar Facet Joints intra-articular injection with Platelet Rich Plasma — Floroscopy guided by C-arm Intraarticular injection in Lumbar facet Joints
  Arms: Group (I) Platelet Rich Plasma
Drug: Lumbar Facet Joints intra-articular injection with a mixture of 0.5% lidocaine and 5mg/ml of betamethasone — Lumbar Facet Joints intra-articular injection
  Arms: Group (II) Corticosteroids

SUMMARY:
Low back pain is an extremely common health problem and recent studies have shown that nearly up to 52% of patients have low back pain caused by lumbar facet joint syndrome. Intra-articular injection of facet joints has gradually become one of the vital therapeutic methods for lumbar facet joint syndrome, Steroid is one of the most commonly used injected drugs; however, previous studies have indicated that it has limited ability in long-term relief of low back pain. Therefore, it seems meaningful to apply a new injectable drug and to prove its effectiveness and safety for the treatment of lumbar facet joint syndrome. Recent studies indicate that autologous platelet rich plasma(PRP) is an appropriate injectable material with great potential in treating many different musculoskeletal disorders and currently it is not yet used on a wide scale as a treatment for lumbar facet joint synovitis. In this study the investigators compare the efficacy and safety of Intra-articular injection of PRP versus conventional steriods in patients with lumbar facet joint synovitis.

DETAILED DESCRIPTION:
The study is conducted upon Thirty patients who present to Ain Shams University hospitals outpatient clinic complaining of chronic low back pain diagnosed to have potential lumbar facet joint syndrome.

Intervention

After taking informed written consent the recruited patients will be subjected to the following:

1. History:

I. Clinical Examination:

1. Full history taking
2. Thorough clinical examination to exclude radicular or neurological manifestation (motor weakness, incontinence, etc.)
3. Analysis of pain using:

   * low back pain visual analogue scale (VAS) at rest: VAS is a subjective numerical pain rating scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain ever experienced.
   * Roland-Morris Disability Questionnaire (RMQ), as experienced by the patient in the last 24 hours, of a total score of 24, where a score of 0 represented no disability and a score of 24 represented the maximum disability .

     * - Oswestry Disability Index (ODI), ODI is currently considered as the gold standard for measuring degree of disability and estimating quality of life in a patient with low back pain. The ODI is comprised of 10 items which reflect the patient's ability to manage their everyday life while dealing with their pain. Each item in the ODI had 6 options to represent a score from 0 to 5, where choice of the first option of the 6 scores 0 and the last scores 5. A percentage score is calculated: total score of the patient/ max score possible x 100%. A 10% change has been identified as being clinically meaningful. The result had 5 levels:
     * minimal disability (0% - 20%)
     * moderate disability (21% - 40%)
     * severe disability (41% - 60%)
     * crippled (61% - 80%)
     * bed-bound or exaggerating symptoms (81% - 100%)(Fairbank et al., 1980). II. Radiological investigation.

Magnetic Resonance Imaging : Done by a single consultant radiologist to detect and grade facet joint synovitis according to the following grading system :

0 : No signal abnormality

1. : Signal abnormality confined to joint capsule
2. : Periarticular signal abnormality involving less than 50 % of the perimeter of the joint*
3. : Periarticular signal abnormality involving more than 50 % of the perimeter of the joint *
4. : Grade 3 with extension of signal abnormality into the intervertebral foramen, ligamentum flavum, pedicle, transverse process, or vertebral body.

   * Signal abnormality may extend into the articular pillar or lamina but does not contribute to the definition of the grade

     * The participants will be randomly assigned for intra-articular injection to either; Group (I) (n =15) to be injected with autologous platelet rich plasma and Group (II) (n=15) to be injected with corticosteroids(a mixture of 0.5% lidocaine and 5mg/ml of betamethasone) . The treated segments will be determined by clinical signs and MRI detected facet joint synovitis .

III. Preparation of Autologous PRP

Under sterile conditions, about 20 ml of peripheral venous blood will be collected with addition of sodium citrate to the test tube. The PRP will be prepared based on the standard 2-step centrifugation method:

1. . The sample is first centrifuged at 1800 rpm for 15 min to separate erythrocytes.
2. Serum supernatant is subjected to the second centrifugation at 3500 rpm for 10 minutes to remove part of the platelet poor plasma and concentrate the platelets.

Finally, approximately 2 to 4 mL of buffy coat autologous PRP is collected in a clear syringe for fluoroscopy guided injection as soon as possible.

IV. Lumbar Facet Joint Injection Injection will be performed under supervision of an experienced pain physician, X-ray guided under fluoroscopy. The site for needle penetration will be marked at the intersection of the beam of a C-arm - a device used to guide the needle to a specific area while watching that needle on a live x-ray screen- and the skin.

Standard antisepsis of the skin will be applied, local anesthesia with 0.5% lidocaine will be administered followed by a 21-G spinal needle insertion into the facet joint space under fluoroscopic control, then the targeted joint will be injected with approximately 0.5 mL of autologous PRP in the first group and with 0.5 to 1 ml of a mixture of 0.5% lidocaine and 5mg/ml of betamethasone in the second group. Multiple joints can be injected in the same setting according to our decision depending on clinical examination and MRI findings.

V. Follow-up and Clinical Evaluation All the patients will be followed at 3 months after the injection and no anti-inflammatory treatment will be given to the patients during the follow up period.

* Clinical evaluation: criteria and scales:

  * low back pain visual analogue scale (VAS) at rest .
  * Roland-Morris Disability Questionnaire (RMQ).
  * Oswestry Disability Index (ODI).
* Magnetic Resonance Imaging For facet joint synovitis detection and grading in the injected joints

Data Management and Analysis:

The collected data is coded, tabulated, and statistically analyzed using SPSS program (Statistical Package for Social Sciences) software version 17.0.

Descriptive statistics will be done for numerical parametric data as mean +/-SD (standard deviation) and minimum & maximum of the range and for numerical non parametric data as median and 1st& 3rd inter-quartile range, while they will be done for categorical data as number and percentage.

Inferential analyses will be done for quantitative variables using independent t-test in cases of two independent groups with parametric data and Mann Whitney U in cases of two independent groups with non parametric data.

Inferential analyses will be done for qualitative data using Chi square test for independent groups. The level of significance will be taken at P value <0.050 is significant, otherwise is non significant. The p-value is a statistical measure for the probability that the results observed in a study could occur by chance.

Ethics:

The study is approved from the Ethical committee of the department of physical medicine , rehabilitation and rheumatology, faculty of medicine, Ain shams university and from the Research Ethical Committee (REC) Ain shams University.

ELIGIBILITY:
Inclusion Criteria:

* • Continuous or intermittent gradually progressive back pain for more than 3 months not significantly improving on medical treatment and/or physical modalities.

  * Patients age between 20 and 40 years.
  * Local / paraspinal pain or tenderness with or without radiation to buttock , groin or thigh.
  * Increase of pain on extension , rotation or lateral bending .
  * MRI detected synovitis of the facet joint as defined and graded by Czervionke and Fenton, 2008.

Exclusion Criteria:

* • Acute low back trauma, fractures, malignancies and inflammatory diseases.

  * Pain score of < 4 at rest on visual analog scale.
  * Radicular neurologic complaints.
  * X-ray findings of long standing facet joint disease as; marked joint space narrowing, subchondral sclerosis or bone deformity/ sponylolithesis.
  * Evident disc herniation by MRI.
  * Prior surgery on the spine.
  * Prior interventional treatment on lumbar facet joints
  * Known hypersenstivity to local anesthesia, corticosteroid, contrast medium or blood derivatives.
  * Local or systemic infection or spinal infection.
  * Uncorrectable coagulopathy
  * Diabetes Mellitus
  * Pregnancy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing total number of lumbar facet joints showing tenderness on palpation on clinical examination | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of total Number of lumbar facet joints showing tenderness on palpation in each participant documented just before the intervention and at 3 month after the intervention
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing maximum active lumber extension angle measured by goniometer | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of Maximum active lumber extension measured by goniometer in each participants documented just before the intervention and at 3 month after the intervention
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing the Visual analogue score (VAS) | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of Visual analogue score documented just before the intervention and at 3 month after the intervention where score of 0 denotes absence of pain and score of 10 denotes maximum pain and decrease in the sore denotes improvement as regards low back pain reported by the participants
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing Roland Morris Disability questionnaire score (RMQ) | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of Roland Morris Disability questionnaire score (RMQ) documented just before the intervention and at 3 month after the intervention, where score 0 denotes absence of any disability and score of 24 denotes maximum disability of the participants and decrease in the score documented denotes improvement
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing Functional questionnaire score - Oswestry Disability Index ODI | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of Oswestry Disability Index score (ODI) documented just before the intervention and at 3 month after the intervention, where score of 0% denotes fully functional participants and score of 100% denotes maximum functional affection and decrease of the score by 10% denotes significant improvement
The Efficacy of lumbar facet joints intra-articular injection of PRP versus conventional Corticosteroids in changing number of lumbar facet joints showing synovitis on MRI and/or improving the grade of severity of the synovitis | at 3 month follow up post intervention for each patient
  In patients complaining of low back pain due to lumbar facet joint disease the investigator asses the efficacy of intra-articular injection of Platelet rich plasma compared to corticosteroids based on comparative analysis of number of lumbar facet joints showing synovitis on MRI and/or improving (decrease in) the grade of severity of the synovitis graded from 0 to 4 according to the extent of lumber facet joint synovitis on MRI documented just before the intervention and at 3 month after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Monir, Professor, Study Director — Faculty of Medicine Ain Shams University; Hala Abdelhady, Professor, Study Director — Faculty of Medicine Ain Shams University; Sahar Fathy, Professor, Study Director — Faculty of Medicine Ain Shams University; Hossam Sakr, Study Director — Faculty of Medicine Ain Shams University; Mohamed Taeimah, MD, Study Director — Faculty of Medicine Ain Shams University; Shahdan Kotb, Principal Investigator — Faculty of Medicine Ain Shams University
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

REFERENCES:
- [Background] Wu J, Du Z, Lv Y, Zhang J, Xiong W, Wang R, Liu R, Zhang G, Liu Q. A New Technique for the Treatment of Lumbar Facet Joint Syndrome Using Intra-articular Injection with Autologous Platelet Rich Plasma. Pain Physician. 2016 Nov-Dec;19(8):617-625. PMID 27906940
- [Background] Wu J, Zhou J, Liu C, Zhang J, Xiong W, Lv Y, Liu R, Wang R, Du Z, Zhang G, Liu Q. A Prospective Study Comparing Platelet-Rich Plasma and Local Anesthetic (LA)/Corticosteroid in Intra-Articular Injection for the Treatment of Lumbar Facet Joint Syndrome. Pain Pract. 2017 Sep;17(7):914-924. doi: 10.1111/papr.12544. Epub 2017 Feb 22. PMID 27989008
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Czervionke LF, Fenton DS. Fat-saturated MR imaging in the detection of inflammatory facet arthropathy (facet synovitis) in the lumbar spine. Pain Med. 2008 May-Jun;9(4):400-6. doi: 10.1111/j.1526-4637.2007.00313.x. PMID 18489631
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Sae-Jung S, Jirarattanaphochai K. Outcomes of lumbar facet syndrome treated with oral diclofenac or methylprednisolone facet injection: a randomized trial. Int Orthop. 2016 Jun;40(6):1091-8. doi: 10.1007/s00264-016-3154-y. Epub 2016 Mar 18. PMID 26987980
- [Background] Zhang J, Middleton KK, Fu FH, Im HJ, Wang JH. HGF mediates the anti-inflammatory effects of PRP on injured tendons. PLoS One. 2013 Jun 28;8(6):e67303. doi: 10.1371/journal.pone.0067303. Print 2013. PMID 23840657
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Maas ET, Juch JN, Ostelo RW, Groeneweg JG, Kallewaard JW, Koes BW, Verhagen AP, Huygen FJ, van Tulder MW. Systematic review of patient history and physical examination to diagnose chronic low back pain originating from the facet joints. Eur J Pain. 2017 Mar;21(3):403-414. doi: 10.1002/ejp.963. Epub 2016 Oct 10. PMID 27723170
- [Background] Manchikanti L, Datta S, Gupta S, Munglani R, Bryce DA, Ward SP, Benyamin RM, Sharma ML, Helm S 2nd, Fellows B, Hirsch JA. A critical review of the American Pain Society clinical practice guidelines for interventional techniques: part 2. Therapeutic interventions. Pain Physician. 2010 Jul-Aug;13(4):E215-64. PMID 20648212
- [Derived] Kotb SY, Sherif NM, Saleh HA, Ahmed SF, Sakr HM, Taeimah MO. The role of intra-articular injection of autologous platelet-rich plasma versus corticosteroids in the treatment of synovitis in lumbar facet joint disease. Saudi Med J. 2022 Nov;43(11):1200-1208. doi: 10.15537/smj.2022.43.11.20220449. PMID 36379530